CLINICAL TRIAL: NCT02581137
Title: M4OC-Prevent: Metformin for Oral Cancer Prevention
Brief Title: Metformin Hydrochloride in Preventing Oral Cancer in Patients With an Oral Premalignant Lesion
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2015-01733; NCI-2015-01733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HHSN2612012000311; N01-CN-2012-00031; 1510157567 (Other: Banner University Medical Center - Tucson); UAZ2015-05-02 (Other: DCP); N01CN00031 (NIH); P30CA023074 (NIH)
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Results first posted 2019-05-23 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Erythroplakia; Hyperplasia; Oral Cavity Carcinoma; Oral Leukoplakia
MeSH Terms: conditions — Erythroplasia; Hyperplasia; Mouth Neoplasms; Leukoplakia, Oral | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prevention (extended-release metformin hydrochloride) (Experimental): Patients receive extended-release metformin hydrochloride PO QD for 2 weeks and then BID for 10-12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Metformin Hydrochloride

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Metformin Hydrochloride — Given PO
  Other Names: APO-Metformin; Cidophage; Dimefor; Glifage; Glucoformin; Glucophage; Glucophage ER; Metformin HCl; Riomet; Siofor

SUMMARY:
This phase IIa trial studies how well metformin hydrochloride works in preventing oral cancer in patients with an oral premalignant lesion (oral leukoplakia or erythroplakia). Oral premalignant lesions look like red or whitish plaques or lesions in the mouth that do not rub off and can be associated with a higher risk of cancer. Metformin hydrochloride may help prevent oral cancer from forming in patients with an oral premalignant lesion.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the clinical response of oral premalignant lesions to 12-14 weeks of metformin (metformin hydrochloride) intervention.

SECONDARY OBJECTIVES:

I. Histologic response to metformin intervention in the target lesion. II. Tissue-based biomarkers: metformin effect on cell proliferation and its molecular targets in the target lesion and in the normal tissue (marker of cell proliferation, Ki67, molecular targets of metformin, including, in order of priority, phosphorylated ribosomal protein S6 kinase [pS6], phosphorylated v-akt murine thymoma viral oncogene homolog 1 [pAKT]S473, phosphorylated eukaryotic translation initiation factor 4E-binding protein 1 [p4EBP], phosphorylated acetyl-CoA carboxylase alpha [pACC]).

III. Tissue-based biomarkers: expression of dysregulated molecular mechanisms and organic cation transporter 3 (OCT 3) in the target lesion and in the normal tissue, including, in order of priority, epidermal growth factor receptor (EGFR), phosphorylated (p)EGFR, tumor protein 53 (p53), phosphatase and tensin homolog (PTEN), phosphorylated mitogen-activated protein kinase 1 (pERK), cyclin-dependent kinase inhibitor 2A (p16), and OCT3.

IV. Tissue-based biomarkers: targeted analysis of cancer-associated genes in the target lesion and blood deoxyribonucleic acid (DNA).

V. Serum and saliva based biomarkers: metformin effect on serum metabolic markers (C-peptide, glycosylated hemoglobin [HbA1c]).

VI. Serum and saliva based biomarkers: metformin concentrations in serum and saliva.

VII Serum and saliva based biomarkers: metformin effect on serum and saliva inflammatory and angiogenic cytokines, including interleukin (IL)-6, IL-8, growth-related oncogene-1 (GRO-1), and vascular endothelial growth factor (VEGF).

EXPLORATORY OBJECTIVES:

I. To characterize changes in the saliva microbiome before and after metformin intervention, including both the absolute microbial load and taxonomic composition.

II. To evaluate the potential microbiome signatures that are correlated with treatment response.

OUTLINE:

Patients receive extended-release metformin hydrochloride orally (PO) once daily (QD) for 2 weeks and then twice daily (BID) for 10-12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants with oral leukoplakia or erythroplakia with mild, moderate, or severe histologic dysplasia, or hyperplasia not associated with mechanical factors such as ill-fitted dentures
* Measurable disease - minimum lesion size of 8 x 3 mm before initial biopsy
* Karnofsky performance status >= 70%
* Leukocytes >= 3,000/microliter
* Absolute neutrophil count >= 1,000/microliter
* Platelets >= 100,000/microliter
* Total bilirubin =< 1.5 × institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =<1.5 × institutional ULN
* eGFR > 40 mL/min using the Cockcroft-Gault equation
* Life expectancy > 3 months
* Willing to use adequate contraception (barrier method, abstinence, subject has had a vasectomy or partner is using effective birth control or is postmenopausal) for the duration of study participation
* Ability to take oral medication
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with diabetes who are taking insulin or oral agents
* History of diabetic ketoacidosis
* Participants may not be receiving any other investigational agents within past 3 months
* History of allergic reactions attributed to compounds of similar chemical composition to metformin or prior use of metformin within the last year
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, human immunodeficiency virus (HIV)-positive, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Oral carcinoma in situ
* History of chronic alcohol use or abuse defined as any one of the following: a) average consumption of 3 or more alcohol containing beverages daily in the past 12 months; b) consumption of 7 or more alcoholic beverages within a 24 hour (hr) period in the past 12 months
* Glycated hemoglobin (HbA1c) > 8%
* Pregnancy or nursing women
* Acute or chronic liver disease, evidence of hepatitis (infectious or autoimmune), cirrhosis or portal hypertension
* History of renal disease
* History of prior head and neck squamous cell carcinoma (HNSCC) unless curatively treated for >= 1 year
* Have received chemotherapy and/or radiation for any malignancy (excluding non-melanoma skin cancer and cancers confined to organs with removal as only treatment) in the past 2 years; ongoing adjuvant hormonal therapy for breast cancer is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-06-10 (Actual); Primary Completion 2017-10-12 (Actual); Study Completion 2025-12-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Lippman, Principal Investigator — The University of Arizona Medical Center-University Campus
Locations (4):
- United States (2):
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
- Canada (2):
  - BC Cancer Research Centre, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia

REFERENCES:
- [Derived] Gutkind JS, Molinolo AA, Wu X, Wang Z, Nachmanson D, Harismendy O, Alexandrov LB, Wuertz BR, Ondrey FG, Laronde D, Rock LD, Rosin M, Coffey C, Butler VD, Bengtson L, Hsu CH, Bauman JE, Hewitt SM, Cohen EE, Chow HS, Lippman SM, Szabo E. Inhibition of mTOR signaling and clinical activity of metformin in oral premalignant lesions. JCI Insight. 2021 Sep 8;6(17):e147096. doi: 10.1172/jci.insight.147096. PMID 34255745

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevention (Extended-release Metformin Hydrochloride)
Started | 26
Completed | 22
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Prevention (Extended-release Metformin Hydrochloride)
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 12
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response to Metformin Intervention
Description: Number of participants with complete and partial clinical response to metformin intervention.
  Criteria for complete and partial clinical response are:
  Complete Response (CR): Disappearance of all evidence of lesion(s). Partial Response (PR): Greater than or equal to 50% reduction in the sum of the products of diameters of lesion(s) measurable at baseline. Non-measurable lesion(s) may not increase greater than or equal to 25% in size and no new lesion may appear.
Time Frame: Baseline to up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Extended-release Metformin Hydrochloride)
Number analyzed (Participants) | 23
Participants | 4

2. Secondary Outcome: Histologic Response to Metformin Intervention
Description: Number of participants with complete and partial histologic response to metformin intervention.
  Criteria for complete and partial histologic response are:
  Complete Response (CR): Complete reversal of dysplasia or hyperplasia to normal epithelium in the target lesion.
  Partial Response (PR): Improvement of the degree of dysplasia or hyperplasia in the target lesion.
Time Frame: Baseline to up to 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prevention (Extended-release Metformin Hydrochloride)
Number analyzed (Participants) | 23
Participants | 14

3. Secondary Outcome: Changes in Cell Proliferation and Its Molecular Targets
Description: Nonparametric methods, e.g. signed rank test, will be performed to evaluate each of the changes in tissue, serum, and saliva markers.
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Changes in Frequent Dysregulated Molecular Mechanisms and OCT Expression
Description: Nonparametric methods, e.g. signed rank test, will be performed to evaluate each of the changes in tissue, serum, and saliva markers. A univariate logistic regression model with the clinical response as the outcome variable will be fitted to explore if any of the expression of frequent dysregulated mechanisms and OCT3 level are associated with the clinical response to metformin hydrochloride.
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Impact of Genomic Alterations on the Biological and Biochemical Consequences and Clinical Response to Metformin Hydrochloride
Description: Nonparametric methods, e.g. signed rank test, will be performed to evaluate each of the changes in tissue, serum, and saliva markers. A univariate logistic regression model with the clinical response as the outcome variable will be fitted to explore if any genomic alterations are associated with the clinical response to metformin hydrochloride.
Time Frame: Up to 14 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Change in Measurements of Metformin Hydrochloride Concentrations in Serum and Saliva
Description: as for outcome 3
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Change in Serum Metabolic Markers
Description: as for outcome 3
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Change in Serum and Saliva Inflammatory and Angiogenic Cytokines
Description: as for outcome 3
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Saliva Microbiome Analyzed Using Flow Cytometry
Description: This will characterize changes in the saliva microbiome before and after metformin intervention, including both the absolute microbial load and taxonomic composition. Will first evaluate changes in alpha diversity among matched pairs using non-parametric analogous Wilcoxon rank-sum test (Mann-Whitney test). To test for significant differences in beta diversity (e.g. if pretreatment and post-treatment samples cluster in principle coordinates analysis space), permutational multivariate analysis of variance (PERMANOVA) will be used.
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Microbiome Signatures Correlated With Treatment Response
Description: Will first evaluate changes in alpha diversity among matched pairs using non-parametric analogous Wilcoxon rank-sum test (Mann-Whitney test). To test for significant differences in beta diversity (e.g. if pretreatment and post-treatment samples cluster in principle coordinates analysis space), PERMANOVA will be used.
Time Frame: Baseline to up to 14 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Prevention (Extended-release Metformin Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 24/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Extended-release Metformin Hydrochloride) (N=26)
oral pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prevention (Extended-release Metformin Hydrochloride) (N=26)
Abdominal pain (Gastrointestinal disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 13
Gastrointestinal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 14
Oral pain (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Upper respiratory infection (Infections and infestations) | 2
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT02581137/Prot_SAP_000.pdf